CLINICAL TRIAL: NCT03117413
Title: Positron Emission Tomography Imaging of Brain Reorganisation of the Central Auditory Cortex in Asymetrical Profound Deaf Patient With a Cochlear Implantation
Acronym: UniTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre de recherche Cerveau et Cognition (CERCO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7797; 2016-A01442-49 (Other: ID-RCB)
Record Dates: First submitted 2017-03-10; First posted 2017-04-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2020-11

CONDITIONS: Profound Hearing Impairment
Keywords: Cochlear implantation; Deafness; Auditory cortex; Auditory plasticity; Tinnitus
MeSH Terms: conditions — Deafness; Tinnitus | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Subjects with asymmetric hearing loss treated with a cochlear implant and a control group of normal hearing subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymmetric hearing loss (Other): Asymmetric hearing loss treated with a cochlear implant will undergo positron emission tomography scan.
  Interventions: Other: Positron emission tomography scan
- Normal hearing subjects (Other): Normal hearing subjects will undergo positron emission tomography scan.
  Interventions: Other: Positron emission tomography scan

INTERVENTIONS:
Other: Positron emission tomography scan — * Binaural hearing assessments: speech recognition in noise and sound source localization
  * Voice perception assessment: voice/non-voice discrimination task, free categorization task
  * Positron emission tomography examinations under ecological auditory stimuli (voice/non-voice discrimination task)

SUMMARY:
Our main objective is to study how the extent of reorganization of the central auditory system is related to the binaural integration in cochlear implanted subjects with asymmetric hearing loss. Subjects with asymmetric hearing loss treated with a cochlear implant and a control group of normal hearing subjects will perform two tests for binaural integration (speech recognition in noise and spatial localization) and two tasks of non-linguistic sounds perception.

DETAILED DESCRIPTION:
Cochlear implantation is the most efficient method to restore hearing in deaf patients. However, about 2/3 of patients have some residual hearing and these patients usually combine two types of auditory information (electrical and acoustical). It is important to know how the brain is processing during two distinct stimulations and how it is related to the auditory level of performance.

Patients and controls will undergo a positron emission tomography scan brain imaging session during a simplified voice/non-voice discrimination task. For each tasks and brain imaging sessions, patients will be stimulated either with the non-implanted ear (acoustical stimulation), the cochlear implant (electrical stimulation) and using both modalities in a binaural condition.

ELIGIBILITY:
Inclusion Criteria:

* cochlear implantation>3 months
* signature of informed consent
* affiliation to social service.

Exclusion Criteria:

* associated neurological disorder
* protected subjects
* epilepsy episodes
* psychotropic medication
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Differences in auditory brain activation between cochlear implanted asymmetric hearing loss subjects and normal hearing subjects in the binaural condition. | Day 1
  Prior to the imaging session, patients performed two human voice interpretation tests. link between temporal activations and performances obtained in binaural integration tasks in the patient group.

SECONDARY OUTCOMES:
differences in auditory brain activation. | Week 3 - Week 5
  Auditory brain activation when the better ear is acoustically stimulated in asymmetric hearing loss subjects and when one ear is stimulated in normal hearing subjects.
Performance level and the pattern of brain activation. | Week 3 - Week 5
  Acoustical or electrical stimulation in asymmetric hearing loss cochlear implanted subjects.
the asymmetry in auditory brain activation for asymmetric hearing loss cochlear implanted subjects. | Week 3 - Week 5
  Electrical and acoustical stimulation will be used.
link between binaural hearing performances and auditory brain activation in the binaural condition. | Week 3 - Week 5
  For the group of cochlear implanted subjects with asymmetric hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, Pr, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, France
  - CERCO, Toulouse, Midi-Pyrénées

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karoui C, James C, Barone P, Bakhos D, Marx M, Macherey O. Searching for the Sound of a Cochlear Implant: Evaluation of Different Vocoder Parameters by Cochlear Implant Users With Single-Sided Deafness. Trends Hear. 2019 Jan-Dec;23:2331216519866029. doi: 10.1177/2331216519866029. PMID 31533581
- [Result] Berland A, Collett E, Gaillard P, Guidetti M, Strelnikov K, Cochard N, Barone P, Deguine O. Categorization of everyday sounds by cochlear implanted children. Sci Rep. 2019 Mar 5;9(1):3532. doi: 10.1038/s41598-019-39991-9. PMID 30837546
- [Result] Strelnikov K, Collett E, Gaillard P, Truy E, Deguine O, Marx M, Barone P. Categorisation of natural sounds at different stages of auditory recovery in cochlear implant adult deaf patients. Hear Res. 2018 Sep;367:182-194. doi: 10.1016/j.heares.2018.06.006. Epub 2018 Jun 12. PMID 29914727